CLINICAL TRIAL: NCT01321437
Title: Phase 2 Study of the Anti-Angiogenesis Agent Axitinib (AG-013736) in Patients With Stage III Malignant Melanoma
Brief Title: Study of the Anti-Angiogenesis Agent Axitinib in Patients With Stage III Malignant Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, John P. Fruehauf, Principal Investigator, University of California, Irvine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCI 10-55 [HS# 2011-8282]; 2011-8282 (Other: University of California, Irvine); WS830279 (Other: Pfizer); NCI-2012-02173 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Melanoma; Malignant Melanoma; Stage IIIA Melanoma; Stage IIIB Melanoma; Stage IIIC Melanoma
Keywords: Melanoma; Axitinib; Anti-angiogenesis; Neoadjuvant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Axitinib (Experimental): Patients receive axitinib PO BID on days 1-28. Treatment repeats every 4 weeks for 2 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery within 14-21 days after completion of treatment. Beginning 28-56 days after surgery, patients receive axitinib PO BID on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity
  Interventions: Procedure: therapeutic conventional surgery; Other: laboratory biomarker analysis; Drug: Axitinib; Other: pharmacological study

INTERVENTIONS:
Procedure: therapeutic conventional surgery — Undergo surgery
Other: laboratory biomarker analysis — Correlative studies
Drug: Axitinib — Axitinib will be administered 5 mg orally twice each day (BID) continuously. Dose adjustments will be based on adverse events.
  Other Names: AG-013736; Inlyta
Other: pharmacological study — Correlative studies

SUMMARY:
The purpose of this research study is to determine the efficacy of Axitinib in treating individuals with Stage III melanoma.

DETAILED DESCRIPTION:
The American Cancer Society estimates that there will be about 68,720 new cases of melanoma (29,900 in men and 25,200 in women) annually in the United States, and about 8,650 people will die from this cancer. The systemic therapy of advanced disease remains palliative until new agents are found that might improve the survival of patients with stage III melanoma.

Melanomas are often vascular, and a decrease in the number of blood vessels that supply the tumor may starve it of needed nutrients. An approach to blocking the growth of blood vessels that supply the tumor is to inhibit the vascular endothelial growth factor receptor tyrosine kinase (VEGFR TK) signaling pathway. Axitinib (AG 013736) is a VEGFR TK inhibitor.

Because of the poor prognosis of patients with stage III melanoma and indications that anti-angiogenesis compounds might have clinically meaningful activity in this disease, a Phase 2 trial of the vascular endothelial growth factor receptor tyrosine kinase (VEGFR TK) inhibitor Axitinib (AG 013736) is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented melanoma with local lymph node stage III metastases.
* No prior systemic therapy. Prior adjuvant therapy with interferon does not count.
* No expectation of further effects of prior anticancer therapy.
* At least 1 target lesion, as defined by RECIST, that has not been irradiated. New lesions that have developed in a previously irradiated field may be used as sites of measurable disease assuming all other criteria are met. All target lesions must have a unidimensional diameter of at least 1 cm for spiral CT scans if the reconstruction algorithm is 0.5 cm), or an standard uptake value (SUV) value ≥ 2.5. Baseline measurements/evaluations must be completed within 4 weeks prior to treatment.
* Adequate bone marrow, hepatic, and renal function documented within 14 days prior to treatment as documented by:

  * absolute neutrophil count (ANC, calculated as the absolute number of neutrophils and bands) ≥1.5 x 10^9 cells/L
  * platelets ≥100 x 10^9 cells /L
  * aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN), unless there are liver metastases in which case AST and ALT ≤5.0 x ULN
  * total bilirubin ≤1.5 x ULN
  * serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥60 mL/min
  * urinary protein <2+ by urine dipstick. If dipstick is ≥2+ then a 24-hour urine collection can be done and the patient may enter only if urinary protein is <2 g per 24 hours
* Age ≥18 years.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* No evidence of preexisting uncontrolled hypertension as documented by 2 baseline blood pressure readings taken at least 1 hour apart. The baseline systolic blood pressure readings must be ≤140, and the baseline diastolic blood pressure readings must be ≤90. Patients whose hypertension is controlled by antihypertensive therapies are eligible.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 7 days prior to treatment.
* Written and voluntary informed consent

Exclusion Criteria:

* Stage IV disease
* History of hemoptysis
* Gastrointestinal abnormalities including:

  * inability to take oral medication
  * requirement for intravenous alimentation
  * prior surgical procedures affecting absorption including gastric resection
  * treatment for active peptic ulcer disease in the past 6 months
  * active gastrointestinal bleeding, unrelated to cancer, as evidenced by hematemesis, hematochezia or melena in the past 3 months without evidence of resolution documented by endoscopy or colonoscopy.
  * malabsorption syndromes.
* Previous treatment with anti-angiogenesis agents including thalidomide, or inhibitors of epidermoid growth factor (EGF), platelet derived growth factor (PDGF), or fibroblast growth factors (FGF) receptors.
* Current use or anticipated inability to avoid use of drugs that are known potent cytochrome P450 3A4 (CYP3A4) inhibitors (ie, grapefruit juice, verapamil, ketoconazole, miconazole, itraconazole, erythromycin, clarithromycin, ergot derivatives, indinavir, saquinavir, ritonavir, nelfinavir, lopinavir, and delavirdine).
* Current use or anticipated inability to avoid use of drugs that are known CYP3A4 or Cytochrome P450 1A2 (CYP1A2) inducers (ie, carbamazepine, dexamethasone, felbamate, omeprazole, phenobarbital, phenytoin, primidone, rifabutin, rifampin, and St. John's wort).
* Active seizure disorder or evidence of brain metastases. (Appropriate imaging should be done to rule out brain metastases.)
* A serious uncontrolled medical disorder or active infection that would impair their ability to receive study treatment.
* History of a malignancy (other than melanoma) except those treated with curative intent for skin cancer (other than melanoma) or in situ breast or cervical cancer or those treated with curative intent for any other cancer with no evidence of disease for 5 years.
* 10. Major surgical procedure or any radiation therapy within 4 weeks of treatment, minimum rest period is 28 days post surgery; maximum rest period 56 days post surgery.
* Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of this protocol.
* Patients (male and female) having procreative potential who are not using adequate contraception or practicing abstinence.
* Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P. Fruehauf, MD, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- Chao Family Comprehensive Cancer Center, Orange, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Axitinib
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Axitinib
Number analyzed (Participants) | 11
Age, Customized [Median (Full Range); unit: years]
  Median Age | 63 [37 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate, Defined as the Percentage of Patients With a Confirmed Clinical Response (CR) or Partial Response (PR)
Description: The response rate (CR or PR according to Response Evaluation Criteria in Solid Tumors (RECIST) will be provided with an exact 95% 2-sided confidence interval calculated using a method based on the F distribution.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 11
Participants | 3

2. Secondary Outcome: Progression-free Survival (PFS)
Description: An estimate of the PFS curve from the Kaplan-Meier method will be presented. Median event time and a 2-sided 95% confidence interval for the median will be provided.
Time Frame: From the date of first dose of axitinib to the first date that criteria for progression were met or the patient died, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib
Number analyzed (Participants) | 11
months | 4 [2.8 to 8.5]

3. Secondary Outcome: Duration of Overall Response
Description: Estimates of duration of overall response from the Kaplan-Meier method will be presented. Median event time (if appropriate) and a 2-sided 95% confidence interval for the median will be provided. The number of CR and PR patients may be small and thereby limit use of the Kaplan-Meier method to provide reliable information. In this case, descriptive statistics or listings will be provided.
Time Frame: From the day the criteria for PR or CR were met to the first day criteria for progression occurred, assessed up to 1 year
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib
Number analyzed (Participants) | 11
months | 8 [3.5 to 13.3]

4. Secondary Outcome: Survival
Description: An estimate of the survival time curve from the Kaplan-Meier method will be presented. Median event time and a 2-sided 95% confidence interval for the median will be provided.
Time Frame: From the day of first dose of axitinib to the day of death, until at least one year after the initial dose for the last treated patient.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib
Number analyzed (Participants) | 11
months | 59 [29.6 to 67.5]

5. Secondary Outcome: Frequencies of Patients Experiencing at Least One Adverse Event (AE)
Description: Will be displayed by body system and preferred term according to Medical Dictionary for Regulatory Activities (MedDRA) terminology. Detailed information collected for each AE will include: description of the event, duration, whether the AE was serious, intensity, relationship to study drug, action taken, and clinical outcome. Intensity (severity) of the AEs will be graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to at least 28 days after the last dose of study drug, on average of 1 year.
Population: Please refer to the Adverse Event tables for specifics.
Measure: Count of Participants; unit: Participants
Arm/Group | Axitinib
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: Adverse events are collected from the time the patient signs the consent from until 28 days after the last administration of the investigational product, on average of 1 year.
Arm/Group | Axitinib
All-Cause Mortality (participants affected / at risk) | 4/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=11)
Hypertension (Blood and lymphatic system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=11)
Hypertension (Blood and lymphatic system disorders) | 5
Proteinuria (Renal and urinary disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Fatigue (General disorders) | 5
Diarrhea (Renal and urinary disorders) | 3
Mucositis (Gastrointestinal disorders) | 3
Hoarseness (General disorders) | 3
Nausea (General disorders) | 3
Weight Loss (General disorders) | 2
Loss of Taste (General disorders) | 2
Pain in Limb (General disorders) | 2
Hypothyroidism (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT01321437/Prot_SAP_000.pdf